CLINICAL TRIAL: NCT03650166
Title: Adoption and Effectiveness of a mHealth Intervention for Hypertension in Older Adults: a Pilot Clinical Trial
Brief Title: High BP and Home Monitoring Experience (HoME) Study
Acronym: HoME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Muldoon, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO18050328
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: High Blood Pressure
Keywords: mhealth; short-messaging system; self-management; home blood pressure monitoring; health literacy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (Active Comparator): Participants receive a personal, validated home BP monitor with oral and written instruction.
  Interventions: Other: Personal BP monitor
- MyBP (Experimental): Participants receive a personal, validated home BP monitor with oral and written instruction. In addition patients receive instruction on, and access to, MyBP. This program provides high BP education through online videos and automated, bidirectional text messaging to assist in continuous home BP self-monitoring.
  Interventions: Other: MyBP; Other: Personal BP monitor

INTERVENTIONS:
Other: MyBP — This program includes online video high BP education and longitudinal, personalized assistance of home BP self-monitoring.
  Arms: MyBP
Other: Personal BP monitor — Battery-powered BP monitor for personal use
  Other Names: A&D Medical Blood Pressure Monitor, model UA-767FAC

SUMMARY:
High blood pressure is a leading risk factor for cardiovascular and kidney disease, yet is uncontrolled in half of affected individuals, and specifically older adults. The investigators have developed an automated program for patient education and personalized assistance of systematic home BP self-monitoring. Reports are sent to primary care providers at regular intervals. This investigation will collect pilot data on feasibility and effectiveness in older adults with and without a caregiver.

DETAILED DESCRIPTION:
Background. Hypertension is a highly prevalent condition and a primary cause of heart disease, kidney failure and cognitive decline. Hypertension is uncontrolled in nearly half of diagnosed adults in the US, with the lowest control rates among older adults (i.e., over 60 y/o). Uncontrolled hypertension is attributable to a mix of factors, most notably suboptimal self-management among patients and clinical inertia due to the reliance on limited BP measurement at office visits, which results in diagnostic uncertainty.

Home BP monitoring (HBPM) is a promising solution to catalyze patient engagement in self-management while offering clinicians reliable and up-to-date data, thereby improving clinical management. Home blood pressure monitoring (HBPM) is now widely recommended as an effective additional tool for improved hypertension management, however broad implementation has not occurred. The convenience of mobile phones has led to high and increasing ownership among all age groups, thus there is great potential to leverage mobile health (mHealth) applications to make HBPM easy, convenient, and even more helpful for both clinicians and patients.

Based upon extensive stakeholder input, the investigators' multidisciplinary team designed a comprehensive mobile phone supported HBPM system called MyBP. MyBP efficiently educates patients via professionally-developed videos and supports bi-weekly BP self-monitoring with recurring feedback using proactive, bidirectional automated texting. Prior pilot testing at three unique clinical sites with middle-aged adults (mean 50 y/o) suggests good usability and positive effects on self-management behaviors. High priority next steps are to: 1) test MyBP specifically with older adults (and caregivers) to fully understand their unique experiences in regards to HBPM via mobile phone, and 2) explore how best to share MyBP data with primary care providers (PCPs). Therefore, the aims of this study are to:

1. Collect pilot data on longitudinal usage of MyBP and BP reduction over 6-9 months within an older adult population.
2. Examine factors influencing adoption and sustained use of MyBP and any associated BP reduction.
3. Identify potentially unique user experiences among older adults with increasing frailty and in those who rely on caregivers.

Methods. Forty-eight older adults (60-85 y/o) with uncontrolled hypertension will be randomized 2:1 to active intervention (MyBP plus a home BP cuff) or usual care (home BP cuff alone) for 6-9 months. Participants will be recruited from UPMC primary care practices. For participants for whom a caregiver has primary responsibility for hypertension-related health behaviors, MyBP will be used by the caregiver. Gait speed will be measured to assess frailty. At baseline and study completion, standardized measurement of home BP will be conducted. Patients and caregivers will complete questionnaires and a semi-structured audio-recorded interview to assess factors associated with MyBP utility and engagement, BP self-management and BP lowering.

Future use of data. Findings will be used to refine the MyBP system design to best fit the target audience and as "preliminary evidence" in an NIH R01 proposal to test in a randomized clinical trial of MyBP in the primary care setting among both mid-life and older adults with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of High blood pressure
* Office systolic BP reading 150 mm Hg or higher
* Owns a cell phone with unlimited texting

Exclusion Criteria:

* Arm circumference > 45 cm
* Dementia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in systolic BP from baseline to trial completion | 5-8 months (Trial duration is not identical across participants but is anticipated to be between 5 and 8 months.)
  Seated BP will be measured in duplicate during each of two baseline assessments (4 total readings) and again in duplicate at each of two assessments at trial completion (4 readings). The primary outcome is the change in average systolic BP from baseline to follow-up. This will be calculated as the average systolic BP at follow-up minus the average systolic BP at baseline. The change in BP in two intervention groups will be compared.

SECONDARY OUTCOMES:
Change in participants' hypertension self-efficacy (confidence in ability to fully understand and manage his or her high BP) | 5-8 months
  Hypertension self-efficacy will be assessed at baseline and trial completion with this question: Please rate your confidence in your ability to fully understand and manage your high BP. [No confidence; A little confidence; Some confidence; High confidence; Very high confidence.] Answers are scored 1-5. Change in score will be compared across the two intervention groups.
Change in systolic BP from baseline to trial mid-point | Approximately 14 weeks
  Seated BP will be measured in duplicate during each of two baseline assessments (4 total readings) and also during two assessments at trial mid-point (4 readings). This secondary outcome is the change in average systolic BP from baseline to trial mid-point. This will be calculated as the average systolic BP at mid-point minus the average systolic BP at baseline. The change in BP in two intervention groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F Muldoon, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Einhorn J, Murphy AR, Rogal SS, Suffoletto B, Irizarry T, Rollman BL, Forman DE, Muldoon MF. Automated Messaging Program to Facilitate Systematic Home Blood Pressure Monitoring: Qualitative Analysis of Provider Interviews. JMIR Cardio. 2023 Dec 4;7:e51316. doi: 10.2196/51316. PMID 38048147